CLINICAL TRIAL: NCT01840865
Title: Impact of Transcranial Slow Oscillating Stimulation on Memory Consolidation During Daytime Slow Wave Sleep in Younger, Healthy Subjects
Brief Title: Effects of Brain Stimulation During Daytime Nap on Memory Consolidation in Younger, Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Agnes Flöel, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nap-tSOS-young
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: young healthy subjects; brain stimulation; tSOS; tDCS; sleep; daytime sleep; nap; memory; memory consolidation
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHAM stimulation (Experimental): SHAM stimulation during periods of Slow Wave Sleep
  Interventions: Device: no stimulation
- 0,75 Hz stimulation (Experimental): slow transcranial oscillating stimulation (~0,75Hz) during periods of Slow Wave Sleep
  Interventions: Device: brain stimulation

INTERVENTIONS:
Device: brain stimulation — oscillating direct current brain stimulation
  Arms: 0,75 Hz stimulation
Device: no stimulation — sham Stimulation
  Arms: SHAM stimulation

SUMMARY:
The beneficial effect of daytime sleep on memory consolidation has been shown in young, healthy subjects. Especially, periods rich in slow-wave sleep (SWS) have shown a memory enhancing effect on hippocampus-dependent declarative memory. Slow oscillatory activity typically occuring during SWS has been implicated in the consolidation effect. In this study we investigate if the consolidation effect can be amplified by the application of a weak transcranial oscillatory electric current within the frequency range of SWS in humans (0,7-0,8 Hz) during daytime SWS.

ELIGIBILITY:
Inclusion Criteria:

* healthy Subjects
* unobtrusive, neuropsychological screening
* age: 18-35 years
* right handed

Exclusion Criteria:

* untreated severe internal or psychiatric diseases
* epilepsy
* other severe neurological diseases eg., previous major stroke, brain tumour
* contraindications to MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Retention of declarative memories after 0.75 Hz stimulation during SWS, vs after sham stimulation during SWS | 4 weeks
  Retention between stimulation conditions (0.75 Hz during SWS, vs sham stimulation during SWS) in the declarative memory task.

SECONDARY OUTCOMES:
Amount of Slow wave Sleep | 4 weeks
  1. Amount of slow wave sleep assessed by standard polysomnographic criteria in 0,75 Hz vs SHAM stimulation during SWS.
2. sleep spindles | 4 weeks
  2. Spindle activity during sleep indicated via several spindle parameters like number, duration, frequency of spindles; compared between 0,75 Hz and SHAM stimulation during SWS.
3. EEG-correlates | 4 weeks
  3. Neuronal correlates (EEG-power in slow oscillation frequency bands induced by 0,75 Hz vs SHAM stimulation during SWS; EEG-correlates of encoding and retrieval of a declarative memory task).
4. further memory systems | 4 weeks
  4. Performance in further memory systems (procedural), compared between 0,75 Hz and SHAM stimulation during SWS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Principal Investigator — Charite Universitätsmedizin Berlin - Neurologie
Locations (1):
- Charite CCM Neurologie Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Mednick SC, Cai DJ, Kanady J, Drummond SP. Comparing the benefits of caffeine, naps and placebo on verbal, motor and perceptual memory. Behav Brain Res. 2008 Nov 3;193(1):79-86. doi: 10.1016/j.bbr.2008.04.028. Epub 2008 May 8. PMID 18554731
- [Background] Mander BA, Santhanam S, Saletin JM, Walker MP. Wake deterioration and sleep restoration of human learning. Curr Biol. 2011 Mar 8;21(5):R183-4. doi: 10.1016/j.cub.2011.01.019. No abstract available. PMID 21377092
- [Background] Mednick S, Nakayama K, Stickgold R. Sleep-dependent learning: a nap is as good as a night. Nat Neurosci. 2003 Jul;6(7):697-8. doi: 10.1038/nn1078. PMID 12819785
- [Derived] Ladenbauer J, Ladenbauer J, Kulzow N, Floel A. Memory-relevant nap sleep physiology in healthy and pathological aging. Sleep. 2021 Jul 9;44(7):zsab002. doi: 10.1093/sleep/zsab002. PMID 33406266